CLINICAL TRIAL: NCT05193357
Title: Home-based Intermittent Pneumatic Compression Therapy: the Impact in Chronic Leg Lymphedema in Patients Treated for Gynecologic Cancer
Brief Title: Home-based Intermittent Pneumatic Compression Therapy for Gynecologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, JiHye Hwang, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: homepump_study
Record Dates: First submitted 2021-12-27; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Gynecologic Cancer; Lymphedema of Leg

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- home-based IPC device (Experimental): Participants used a device produced by Maxstar Corp. (Gimpo, South Korea), which specializes in pneumatic compression appliance manufacture. The IPC device (UAM-9306NB) was cleared by National Institute of Medical Device Safety Information (NIDS) of Korea (approval number: 18-4745). This device consists of a six-chamber pneumatic sleeve and a gradient-sequential pneumatic pump.
  Interventions: Device: home-based intermittent pneumatic compression (IPC) device

INTERVENTIONS:
Device: home-based intermittent pneumatic compression (IPC) device — During the intervention, two programmed modes were used. The first mode, which mimics the MLD massage technique, begins with the inflation of the proximal chamber. After reaching the target pressure, the next chamber consecutively inflates while the initially inflated proximal chamber deflates. The inflation time of each chamber is 3 seconds with holding time of 1 second. The deflation and resting time of each chamber is 7 seconds (pressure setting: 40-60 mmHg). After 30 minutes of the first mode, the second mode, which is the conventional mode of sequential inflation from distal to proximal chambers while sustaining the pressure of the previously inflated chambers, was applied for 30 minutes (pressure setting: 80-100 mmHg, inflation time of each chamber: 6 seconds, holding time: 1 second, deflation time of each chamber: 7 seconds). Participants were instructed to use the IPC device with that 1-hour cycle twice a day for four weeks.

SUMMARY:
Investigators conducted a prospective study of cancer patients to investigate the efficacy, quality of life, satisfaction, and safety of a home-based intermittent pneumatic compression (IPC) device during the maintenance phase of lower extremity lymphedema. This device has a unique mode designed to mimic the manual lymphatic drainage (MLD) technique and thereby gently facilitate lymphatic draining of proximal extremities.

ELIGIBILITY:
Inclusion Criteria:

* stage 3 chronic unilateral secondary leg lymphedema
* aged 20-70 years
* underwent 1-2 cycle of treatment of decongestive phase with current inter-limb volume difference of more than 10%
* stable limb-volume change (within 10%) during the preceding 3 months
* capacity for self-maintenance care for lymphedema (multilayer limb bandaging, compression garments, and MLD)

Exclusion Criteria:

* bilateral leg lymphedema
* current cancer metastasis
* ongoing chemotherapy or radiation therapy
* acute inflammation
* venous thrombosis, or chronic venous insufficiency
* systemic etiologies of edema
* congestive heart failure
* patients taking medication that influenced body fluid or electrolytes

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Change of Inter-limb volume difference ratio | Baseline, after 1 month (4-week)
  Investigators measured three leg volumes: the distal leg volume (distal volume: from the smallest circumference at the ankle (B-measure) to the calf circumference right below the knee bend (D-measure)), the whole leg volume (limb volume without the foot up to the mid-thigh region (F-measure)), and the proximal leg volume (subtraction of the distal leg volume from the whole leg volume)

SECONDARY OUTCOMES:
Change of Quality of life (Lymph-ICF-LL) | Baseline, after 1 month (4-week)
  Lymphedema Functioning, Disability, and Health Questionnaire for Lower Limb Lymphedema (Lymph-ICF-LL).
  Questionnaire contains 28 questions divided into 5 domains: physical function, mental function, general tasks/household activities, mobility activities, and life domains/social life. Each question is scored from 0 (not at all) to 10 (a lot), with lower scores representing better QOL. The total scores and 5 domain scores were calculated by summation.
Participant satisfaction questionnaire | after 1 month (4-week)
  The questionnaire contained 6 items related to the subjective effects of the IPC device related to volume reduction, pain, heaviness, skin hardness, ease of use, and overall satisfaction with the home therapy offered by the device. Each question was answered using a 5-point scale from 1 (not at all) to 5 (very much).

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No